CLINICAL TRIAL: NCT03094390
Title: The Impact of Thoracic Fluid Content Measured by Cardiometry on Prediction of Failure of Weaning From Mechanical Ventilation
Brief Title: Thoracic Fluid Content in Prediction of Failure of Weaning From Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Principal investigator, Lecturer of anesthesia and critical care medicine, Cairo University
Other Study IDs: N-18-2017
Record Dates: First submitted 2017-03-20; First posted 2017-03-29 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Mechanical Ventilation Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to test the accuracy of the total thoracic fluid content (TFC) measured by cardiometry can predict weaning failure. Area under receiver operating characteristic curve (AUROC) will be determined, sensitivity, specificity, and best cutoff value will be calculated for TFC in prediction of weaning failure.

DETAILED DESCRIPTION:
Weaning from mechanical ventilation is a serious and challenging process in critical care practice. Weaning failure is associated with poor patient outcomes. Increased mortality in patients with failed weaning was due to development of complications related to re-intubation. Detection and correction of the cause of failed spontaneous breathing trial (SBT) helps the intensives to improve the outcome of the next trials.

Fluid overload and positive cumulative fluid balance is a risk factor of weaning failure in both cardiac and non-cardiac patients.

Many tools for prediction of lung congestion as a risk factor for weaning failure have been reported. The gold standard for detection of cardiac cause of weaning failure was pulmonary artery catheter. More simple tools had been investigated for detection of cardiac cause of weaning failure in patients with or without previous cardiac dysfunction such as extravascular lung water and B-natriuretic peptide (BNP) levels.

Although measurement of extravascular lung water is a reliable tool for prediction of cardiac cause of weaning failure, it has the disadvantage of the need of advanced monitor with invasive arterial line. Bioreactance is a new technology used for measurement of cardiac output and total thoracic fluid content (TFC). More recently, electrical velocimetry is a newer technology with good performance in cardiac output monitoring. The use of electrical velocimetry in measurement of TFC has the advantage of being non-invasive with no need for advanced skills. The aim of this work is to validate the use of TFC (measured by electrical velocimetry) in prediction of weaning outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or more scheduled for a spontaneous weaning trial (SBT) on pressure support ventilation.

Exclusion Criteria:

* Age < 18 years old.
* Pregnant patients.
* Neuromuscular disease (stroke, myasthenia gravis and Guillain-Barrésyndrome).
* Tracheostomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or more scheduled for a spontaneous weaning trial (SBT) using pressure support ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Total thoracic fluid content (TFC) | 5 minutes before spontaneous breathing trial
  the value of TFC measured by cardiometry device (in liters)

SECONDARY OUTCOMES:
rapid shallow breathing index | 5 minutes before spontaneous breathing trial.
  the respiratory rate divided by the tidal volume (in liters)
P/F ratio | 5 minutes before spontaneous breathing trial and 5 minutes before patient extubation
  pressure of arterial oxygen (in mmHg) divided by fraction of inspired oxygen
fluid balance | during the last 24 hours before the weaning trial
  the total fluid intake minus the fluid output (in liters)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mukhtar, Professor, Study Director — Head of research committee section in anesthesia department
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No